CLINICAL TRIAL: NCT00254163
Title: A Prospective, Randomized, Open Label, Phase III Trial of Fludarabine, Cyclophosphamide, and Rituximab vs. Pentostatin, Cyclophosphamide, and Rituximab in Previously Untreated or Treated B-cell Chronic Lymphocytic Leukemia
Brief Title: Fludarabine, Cyclophosphamide, and Rituximab Versus Pentostatin, Cyclophosphamide, and Rituximab in Previously Untreated or Treated B-Cell Chronic Lymphocytic Leukemia Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: US Oncology Research (Industry)
Collaborators: Astex Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 03017; NIP-03-007 (Other: Hospira)
Record Dates: First submitted 2005-11-09; First posted 2005-11-15 (Estimated); Results first posted 2016-11-03 (Estimated); Last update posted 2016-11-03 (Estimated); Status verified 2016-09

CONDITIONS: B-Cell Chronic Lymphocytic Leukemia
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell | interventions — fludarabine; Cyclophosphamide; Rituximab; Pentostatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Fludarabine, Cyclophosphamide, and Rituximab (Active Comparator): Fludarabine, Cyclophosphamide, and Rituximab (dosage based on day in cycle)
  Interventions: Drug: Fludarabine; Drug: Cyclophosphamide; Drug: Rituximab
- Pentostatin, Cyclophosphamide, and Rituximab (Experimental): Pentostatin, Cyclophosphamide, and Rituximab (dosage depends on day in cycle)
  Interventions: Drug: Cyclophosphamide; Drug: Rituximab; Drug: Pentostatin

INTERVENTIONS:
Drug: Fludarabine
  Arms: Fludarabine, Cyclophosphamide, and Rituximab
Drug: Cyclophosphamide
Drug: Rituximab
Drug: Pentostatin
  Other Names: Nipent
  Arms: Pentostatin, Cyclophosphamide, and Rituximab

SUMMARY:
The purpose of this research study is to find out what effects (good and bad) the combination of Nipent+Cytoxan+Rituxan has on CLL cancer compared to Fludara+Cytoxan+Rituxan. While all of these drugs are approved by the Food and Drug Administration (FDA) for the treatment of other cancers, these combinations are experimental for the treatment of CLL.

ELIGIBILITY:
INCLUSION CRITERIA:

Patients will be eligible for inclusion in this study if they meet all of the following criteria:

* Progressive, histologically proven B-cell CLL.
* Stage II, III, or IV B-cell CLL, as defined by Appendix III.

Note: The pathology or flow cytometry (of peripheral blood or a bone marrow) report, done by the local laboratory which documents these findings, must be included in the source documents. The SI must review the above pathology report or flow cytometry report results (including bone marrow aspirate analysis and CD5 and CD20 results) by fax, prior to registration, to confirm each patient's eligibility. Results should be consistent with typical B-cell CLL. If Dr. Reynolds is not available to review these documents, they must be reviewed by Dr. Nicholas J. Di Bella.

* Patient must be CD20 +
* Patient must be CD5+ (CD5 >70%)
* No more than 1 prior course (regimen) of chemotherapy, which can include Fludara or Rituxan
* No prior radiation therapy, except for the treatment of skin cancer or a nonmalignant condition.
* If patient has lymph node involvement, a CT scan confirming measurable tumor size (lymph node must be >1 cm in its longest transverse diameter).
* SI has been notified IF patient is on replacement steroids at time of registration.
* Age greater than 18 years.
* ECOG performance status of 0-2 (Appendix I).
* Normal renal function (creatinine <1.5 mg/dL and BUN <25 mg/dL).
* Absolute neutrophil count (ANC) greater than 1,000 cells/µL, platelet count greater than 50,000 cells/µL, and hemoglobin greater than 9 g/dL.
* Bilirubin less than 2.0 mg/dL, and AST and ALT less than 5 times the upper limit of normal.
* Negative serum pregnancy test within 7 days prior to registration (female patients of childbearing potential).
* Agrees to use an acceptable method of birth control, if fertile patient (male or female), to avoid pregnancy for the duration of the study and for at least 3 months thereafter.
* A signed Patient Informed Consent Form has been obtained.
* A signed Patient Authorization Form has been obtained.

EXCLUSION CRITERIA:

Patients will be excluded from this study if they meet any of the following criteria:

* Any disease other than histologically confirmed progressive, Stage II, III, or IV CLL.
* Well differentiated lymphocytic lymphoma in nodes without lymphocytosis.
* More than 1 prior course (regimen) of chemotherapy.
* Any radiation for the treatment of CLL.
* Any prior Nipent.
* Known to be CD20 negative (CD20 <20%).
* Pregnant or lactating, or has a positive pregnancy test.
* Has a history of other malignancy (other than in situ cervical cancer, carcinoma intraepithelial neoplasia, or non-melanoma skin cancer) within the last 5 years, which could affect the administration of these study drugs or assessment of current CLL.
* Known to be HIV positive.
* Uncontrolled thyroid disease or uncontrolled abnormal thyroid function.

Note: Patients with thyroid disease that is controlled with medication may participate.

* A history of recent, unstable organic heart disease or stable organic heart disease with LVEF <50%.
* A known hypersensitivity to Fludara, Nipent, Rituxan, or Cytoxan, or any component of these drugs.
* Autoimmune hemolytic anemia.
* Unable to comply with requirements of study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 184 (Actual)
Dates: Start 2003-12; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Craig Reynolds, MD, Principal Investigator — US Oncology Research
Locations (11):
- United States (11):
  - Cancer Centers of Florida, P.A., Ocoee, Florida
  - Hope Center, Terre Haute, Indiana
  - Alliance Hematology Oncology PA, Westminster, Maryland
  - St Joseph Oncology, Inc, Saint Joseph, Missouri
  - New York Oncology Hematology, PC, Albany, New York
  - Northwestern Carolina Oncology Hemato, Hickory, North Carolina
  - Medical Oncology Associates, Kingston, Pennsylvania
  - South Texas Cancer Center-McAllen, McAllen, Texas
  - Texas Oncology Cancer Center-Sugar Land, Sugar Land, Texas
  - Cancer Care Northwest-South, Spokane, Washington
  - Yakima Valley Mem Hosp/North Star Lodge, Yakima, Washington

RESULTS

PARTICIPANT FLOW:
Groups:
- FCR Arm: Fludarabine, Cyclophosphamide, and Rituximab
- PCR Arm: Pentostatin, Cyclophosphamide, and Rituximab
Period: Overall Study
Arm/Group | FCR Arm | PCR Arm
Started | 92 | 92
Completed | 47 | 46
Not Completed | 45 | 46
Not completed — Adverse Event | 29 | 26
Not completed — Patient request/withdrew consent | 6 | 4
Not completed — Investigator request | 1 | 3
Not completed — Failed entry | 1 | 3
Not completed — Progressive disease | 0 | 1
Not completed — Death | 0 | 1
Not completed — Other | 8 | 8

BASELINE CHARACTERISTICS:
Population: ITT population
Groups:
- Total: Total of all reporting groups
Arm/Group | FCR Arm | PCR Arm | Total
Number analyzed (Participants) | 92 | 92 | 184
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.3 (10.2) | 63.6 (9.9) | 63.5 (10.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27 | 22 | 49
  Male | 65 | 70 | 135
Race/Ethnicity, Customized [Number; unit: participants]
  Caucasion | 81 | 84 | 165
  Black | 7 | 5 | 12
  Hispanic | 2 | 3 | 5
  Mixed: Black/Indian | 2 | 0 | 2
Region of Enrollment [Number; unit: participants]
  United States | 92 | 92 | 184

OUTCOME MEASURES:

1. Primary Outcome: Infection Rate
Description: infection=febrile events requiring treatment
Time Frame: 6 cycles of 28-day for FCR and 8 cycles of 21-day for PCR, or until PD, CR, or intolerable toxicity
Population: Per protocol population
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | FCR Arm | PCR Arm
Number analyzed (Participants) | 86 | 85
percentage of participants | 31.4 [21.8 to 42.3] | 36.5 [26.3 to 47.6]

2. Secondary Outcome: Infective Event Rate
Description: infective events=temperature >101 without symptoms or temp <101 with symptoms
Time Frame: 6 cycles of 28-day for FCR and 8 cycles of 21-day for PCR, or until PD, CR, or intolerable toxicity
Population: Per protocol population
Measure: Number; unit: percentage of infective events
Arm/Group | FCR Arm | PCR Arm
Number analyzed (Participants) | 86 | 85
percentage of infective events | 38 | 45

3. Secondary Outcome: Percentage of Patients Hospitalized
Description: Percentage of patients who were hospitalized due to any reasons during the study period.
Time Frame: 6 cycles of 28-day for FCR and 8 cycles of 21-day for PCR, or until PD, CR, or intolerable toxicity
Population: Per protocol population
Measure: Number; unit: percentage of participants
Arm/Group | FCR Arm | PCR Arm
Number analyzed (Participants) | 86 | 85
percentage of participants | 35 | 43.5

4. Secondary Outcome: Hematologic Recovery
Description: defined as Hb >11g/dL and a platelet count >100 × 10^3/mm^3
Time Frame: 2 months post-treatment
Population: Per protocol population
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | FCR Arm | PCR Arm
Number analyzed (Participants) | 86 | 85
percentage of participants | 3.5 [0.7 to 9.9] | 14.1 [7.5 to 23.4]

5. Secondary Outcome: Mean Absolute Neutrophil Count (ANC) at Post-treatment
Description: mean Absolute Neutrophil Count (ANC) measured 2 months (8-10 weeks) following the last dose of study treatment
Time Frame: 2 months post-treatment
Population: Per protocol population
Measure: Mean (Standard Deviation); unit: 10^3 cells/mm^3
Arm/Group | FCR Arm | PCR Arm
Number analyzed (Participants) | 86 | 85
10^3 cells/mm^3 | 1.7 (0.9) | 2.2 (1.6)

6. Secondary Outcome: Complete Remission (CR)
Description: Definitions of response is evaluated using guidelines proposed by the National Cancer Institute-Sponsored Working Group for Chronic Lymphocytic Leukemia.
  Complete remission (CR) requires all of the following for a period of at least 2 months:
  1. Absence of lymphadenopathy by physical examination and appropriate radiographic techniques. Lymph nodes must be <1 cm.
  2. No evidence of hepatomegaly or splenomegaly.
  3. Absence of constitutional symptoms.
  4. Normal CBC as exhibited by:
     * Polymorphonuclear leukocytes ≥ 1,500/mm^3
     * Platelets > 100,000/mm^3
     * Hemoglobin > 11.0 g/dL (untransfused)
  5. Bone marrow aspirate and biopsy should be performed 2 months after clinical and laboratory results demonstrate that all of the requirements listed in 1-4 have been met to demonstrate that a CR has been achieved. The marrow sample must be at least normocellular for age, with less than 30% of the nucleated cells being lymphocytes.
  Lymphoid nodules should be absent.
Time Frame: 6 cycles of 28-day for FCR and 8 cycles of 21-day for PCR, or until PD, CR, or intolerable toxicity
Population: Per protocol population
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | FCR Arm | PCR Arm
Number analyzed (Participants) | 86 | 85
percentage of participants | 14.0 [7.4 to 23.1] | 7.1 [2.6 to 14.7]

7. Secondary Outcome: Objective Remission Rate (ORR)
Description: Complete remission (CR) see Outcome Measure 6. Partial remission (PR) must exhibit criteria 1 and 2 as well as one or more of the remaining features for at least 2 months.
  1. ≥50% decrease in peripheral blood lymphocyte count from the pretreatment baseline value.
  2. ≥50% reduction in lymphadenopathy.
  3. ≥50% reduction in the size of the liver and/or spleen.
  4. Polymorphonuclear leukocytes ≥ 1,500/mm^3 or 50% improvement over baseline.
  5. Platelets >100,000/mm^3 or 50% improvement over baseline.
  6. Hemoglobin >11.0 g/dL or 50% improvement over baseline without transfusions. Nodular partial remission (nPR) is defined as a CR with persistent bone marrow nodules; Objective Remission (OR) = CR + PR + nPR.
Time Frame: 6 cycles of 28-day for FCR and 8 cycles of 21-day for PCR, or until PD, CR, or intolerable toxicity
Population: Per protocol population
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | FCR Arm | PCR Arm
Number analyzed (Participants) | 86 | 85
percentage of participants | 59.3 [48.2 to 69.8] | 49.4 [38.4 to 60.5]

8. Secondary Outcome: Progression-free Survival (PFS) Rate at 1-year
Description: PFS is measured from the date of randomization to the date of first documented disease progression or date of death, whichever comes first. If a patient neither progresses nor dies, this patient will be censored at last contact date
Time Frame: 12 months after registered.
Population: Per protocol population
Measure: Number (95% Confidence Interval); unit: probability of Progression-free Survival
Arm/Group | FCR Arm | PCR Arm
Number analyzed (Participants) | 86 | 85
probability of Progression-free Survival | 0.86 [0.76 to 0.92] | 0.84 [0.74 to 0.90]

9. Secondary Outcome: Progression-free Survival (PFS) Rate at 2-year
Description: as for outcome 8
Time Frame: 24 months after registered.
Population: Per protocol population
Measure: Number (95% Confidence Interval); unit: Probability of Progression-free Survival
Arm/Group | FCR Arm | PCR Arm
Number analyzed (Participants) | 86 | 85
Probability of Progression-free Survival | 0.72 [0.60 to 0.81] | 0.63 [0.51 to 0.73]

ADVERSE EVENTS:
Time Frame: During the whole treatment period, up to 30 days following last dose.
Description: The safety population, which received at least one of study treatment, was included in the analysis of adverse event. Patients included in this study were 88 and 89 in FCR arm and PCR arm, respectively.
Arm/Group | FCR Arm | PCR Arm
Serious Adverse Events (participants affected / at risk) | 18/88 | 22/89
Other Adverse Events (participants affected / at risk) | 86/88 | 87/89
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | FCR Arm (N=88) | PCR Arm (N=89)
ABDO ENLARGE (Gastrointestinal disorders) | 1 (1) | 0 (0)
ACIDOSIS (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
ALLERG REACT (Immune system disorders) | 1 (1) | 0 (0)
ANEMIA (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
CARDIOVASC DIS (Cardiac disorders) | 0 (0) | 1 (1)
CELLULITIS (Infections and infestations) | 1 (1) | 0 (0)
COLITIS (Gastrointestinal disorders) | 0 (0) | 1 (1)
CHEST PAIN (General disorders) | 0 (0) | 2 (2)
CONFUS (General disorders) | 0 (0) | 1 (1)
COUGH INC (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
DEHYDRAT (Gastrointestinal disorders) | 0 (0) | 3 (3)
DIARRHEA (Gastrointestinal disorders) | 1 (1) | 0 (0)
DYSPNEA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 4 (4)
EDEMA (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
EDEMA LUNG (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
EFFUS PLEURAL (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
FEBRILE NEUTROPENIA (Blood and lymphatic system disorders) | 5 (5) | 5 (5)
FEVER (General disorders) | 6 (7) | 5 (7)
HEART FAIL RIGHT (Cardiac disorders) | 0 (0) | 1 (1)
HYPOXIA (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
IMMUNOGLOBUL DEC (Immune system disorders) | 1 (1) | 0 (0)
INFECT (Infections and infestations) | 1 (1) | 2 (2)
KIDNEY FAIL (Renal and urinary disorders) | 0 (0) | 3 (3)
LIVER FAIL (Hepatobiliary disorders) | 0 (0) | 1 (1)
LUNG DIS (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0)
MYASTHENIA (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
NEUTROPENIA (Blood and lymphatic system disorders) | 4 (4) | 4 (4)
PAIN (General disorders) | 0 (0) | 1 (2)
PAIN ABDO (Gastrointestinal disorders) | 0 (0) | 1 (1)
PANCYTOPENIA (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
PNEUMONIA (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2)
RESPIRAT DIS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
SEPSIS (Infections and infestations) | 2 (2) | 2 (2)
SINUSITIS (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
STOMATITIS (Gastrointestinal disorders) | 1 (1) | 0 (0)
TACHYCARDIA (Cardiac disorders) | 0 (0) | 1 (1)
TUMOR LYSIS SYNDROME (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
VOMIT (Gastrointestinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | FCR Arm (N=88) | PCR Arm (N=89)
ALLERG REACT (Immune system disorders) | 2 (2) | 6 (7)
ALOPECIA (Skin and subcutaneous tissue disorders) | 4 (4) | 6 (6)
ANEMIA (Blood and lymphatic system disorders) | 45 (126) | 34 (82)
ANOREXIA (Gastrointestinal disorders) | 14 (20) | 23 (31)
ANXIETY (Nervous system disorders) | 2 (2) | 5 (5)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 3 (3) | 7 (8)
ASTHENIA (General disorders) | 48 (99) | 53 (97)
BILIRUBINEM (Metabolism and nutrition disorders) | 6 (7) | 2 (2)
CHILLS (General disorders) | 18 (21) | 16 (25)
CONSTIP (Gastrointestinal disorders) | 16 (21) | 9 (16)
COUGH INC (Respiratory, thoracic and mediastinal disorders) | 8 (9) | 10 (11)
CREATININE INC (Metabolism and nutrition disorders) | 3 (3) | 7 (10)
DEHYDRAT (Gastrointestinal disorders) | 2 (2) | 5 (6)
DIARRHEA (Gastrointestinal disorders) | 13 (18) | 12 (16)
DIZZINESS (Nervous system disorders) | 7 (8) | 7 (8)
DYSPEPSIA (Gastrointestinal disorders) | 9 (16) | 3 (3)
DYSPNEA (Respiratory, thoracic and mediastinal disorders) | 9 (9) | 7 (9)
EDEMA (Blood and lymphatic system disorders) | 3 (3) | 8 (14)
EDEMA PERIPH (Blood and lymphatic system disorders) | 6 (6) | 5 (5)
FEVER (General disorders) | 18 (24) | 30 (45)
HEADACHE (General disorders) | 10 (15) | 4 (5)
HYPERGLYCEM (Metabolism and nutrition disorders) | 6 (8) | 6 (7)
INFECT (Infections and infestations) | 5 (8) | 5 (7)
INSOMNIA (General disorders) | 8 (10) | 3 (4)
LDH INC (Metabolism and nutrition disorders) | 5 (5) | 5 (7)
LEUKOPENIA (Blood and lymphatic system disorders) | 41 (267) | 34 (135)
NAUSEA (Gastrointestinal disorders) | 47 (81) | 49 (123)
NEUROPATHY (Nervous system disorders) | 3 (3) | 6 (10)
NEUTROPENIA (Blood and lymphatic system disorders) | 72 (271) | 68 (185)
PAIN (General disorders) | 6 (7) | 9 (11)
PAIN ABDO (Gastrointestinal disorders) | 6 (7) | 5 (9)
RASH (Skin and subcutaneous tissue disorders) | 11 (16) | 12 (20)
SGOT INC (Metabolism and nutrition disorders) | 6 (6) | 3 (3)
SGPT INC (Metabolism and nutrition disorders) | 9 (9) | 2 (2)
SKIN DRY (Skin and subcutaneous tissue disorders) | 5 (6) | 6 (6)
STOMATITIS (Gastrointestinal disorders) | 7 (11) | 4 (4)
TASTE PERVERS (Gastrointestinal disorders) | 7 (9) | 10 (11)
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 33 (87) | 24 (44)
URIN FREQUENCY (Renal and urinary disorders) | 6 (6) | 2 (2)
VOMIT (Gastrointestinal disorders) | 14 (18) | 25 (44)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No